CLINICAL TRIAL: NCT00948935
Title: Phase II Combination of Gemcitabine (Fixed Dose-rate Infusion, FDR), Irinotecan and Panitumumab in Patients With Advanced and Metastatic Biliary Tract Adenocarcinoma
Brief Title: Study of Gemcitabine, Irinotecan and Panitumumab in Patients With Advanced and Metastatic Biliary Tract Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06208
Record Dates: First submitted 2009-05-15; First posted 2009-07-29 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Biliary Cancer; Cholangiocarcinoma
Keywords: Biliary Cancer; Cholangiocarcinoma; Panitumumab
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Irinotecan; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Gemcitabine (Days 1, 8), irinotecan (days 1, 8) and panitumumab (day 1) every 3 weeks as a cycle. Continue until disease progression or unacceptable toxicities.
  Interventions: Drug: Gemcitabine, Irinotecan, Panitumumab

INTERVENTIONS:
Drug: Gemcitabine, Irinotecan, Panitumumab — Gemcitabine 1000 mg/m2 over 100 minutes(Days 1, 8), irinotecan 100 mg/m2 IV over 60 minutes(days 1, 8) and panitumumab 9 mg/kg IV (day 1) every 3 weeks as a cycle. Continue until disease progression or unacceptable toxicities.

SUMMARY:
This study evaluates the combination chemotherapy with gemcitabine, irinotecan and panitumumab in patients with advanced biliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed local advanced unresectable/metastatic adenocarcinoma of biliary tract
* measurable disease
* available tumor tissue for investigational immunohistochemical evaluations
* ECOG PS 0-2
* No prior chemotherapy, biologic therapy or radiation therapy
* Age Eighteen and older
* Lab values per protocol

Exclusion Criteria:

* Life expectancy less than three months
* Concurrent use of chemotherapy not indicated in the study protocol or any other investigational agents and patients who have received investigational drugs less than four weeks prior to enrollment
* Prior therapy, which affects or targets the EGF pathway
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer
* Recovery from major surgery within three weeks of the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Giantonia, MD, Principal Investigator — Abramson CC
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sohal DP, Mykulowycz K, Uehara T, Teitelbaum UR, Damjanov N, Giantonio BJ, Carberry M, Wissel P, Jacobs-Small M, O'Dwyer PJ, Sepulveda A, Sun W. A phase II trial of gemcitabine, irinotecan and panitumumab in advanced cholangiocarcinoma. Ann Oncol. 2013 Dec;24(12):3061-5. doi: 10.1093/annonc/mdt416. Epub 2013 Oct 20. PMID 24146220

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at Five Months
Time Frame: 5 months
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 35
percentage of participants | 69

2. Secondary Outcome: Response Rate From Combination Chemotherapy
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 35
Participants
  Complete Response | 2
  Partial Response | 9
  Stable Disease | 15
  Progressive Disease | 2
  Not Assessable | 7

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 21/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=35)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (5)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Free Air (Gastrointestinal disorders) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 3 (5)
Abdomen NOS (Infections and infestations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Neurological Meningitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chronic obstructive pulmonary disease (Reproductive system and breast disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Peripheral arterial ischemia (Vascular disorders) | 1 (2)
Thrombosis/thombus/embolism (Vascular disorders) | 4 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=35)
bloating (Gastrointestinal disorders) | 5 (5)
abdominal cramping (Gastrointestinal disorders) | 1 (2)
abdominal fullness (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 16 (18)
acidosis (Metabolism and nutrition disorders) | 1 (1)
acne-form (Skin and subcutaneous tissue disorders) | 2 (2)
acute arterial occulsion LLE (Vascular disorders) | 1 (1)
infusion reaction (General disorders) | 3 (3)
acute renal failure (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 28 (107)
alkaline phosphatase (high) (Metabolism and nutrition disorders) | 22 (59)
alkalosis (Metabolism and nutrition disorders) | 1 (1)
allergic rhinitis (Immune system disorders) | 1 (1)
tape allergy (Immune system disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 19 (20)
Alanine Aminotransferase (high) (Metabolism and nutrition disorders) | 16 (35)
amylase (high) (Metabolism and nutrition disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 20 (90)
anorexia (Gastrointestinal disorders) | 13 (17)
anxiety (Psychiatric disorders) | 9 (10)
ascending cholangitis (Infections and infestations) | 1 (1)
ascites (Gastrointestinal disorders) | 4 (4)
Aspartate Aminotransferase (high) (Metabolism and nutrition disorders) | 24 (55)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
edema (Blood and lymphatic system disorders) | 17 (42)
back pain (Musculoskeletal and connective tissue disorders) | 12 (22)
belching (Gastrointestinal disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 11 (14)
bilirubin (high) (Metabolism and nutrition disorders) | 17 (32)
hemorrhoids (Vascular disorders) | 1 (1)
blurred vision (Eye disorders) | 3 (3)
Body Aches (Musculoskeletal and connective tissue disorders) | 1 (1)
low calcium (Metabolism and nutrition disorders) | 28 (94)
high calcium (Metabolism and nutrition disorders) | 2 (3)
cellulitis (Infections and infestations) | 1 (1)
cerebro-vascular ischemia (Nervous system disorders) | 1 (1)
cheliosis (Skin and subcutaneous tissue disorders) | 3 (3)
Chills (General disorders) | 4 (6)
cold (respiratory) (Immune system disorders) | 1 (1)
confusion (Psychiatric disorders) | 3 (3)
congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
conjuctivitis (Infections and infestations) | 3 (5)
constipation (Gastrointestinal disorders) | 23 (33)
contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 13 (17)
high creatinine (Metabolism and nutrition disorders) | 7 (8)
decreased appetite (Gastrointestinal disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 13 (17)
dementia (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 8 (14)
dermal changes (Blood and lymphatic system disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 25 (51)
dizziness (General disorders) | 12 (17)
dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
dry eye (Eye disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 3 (4)
dry skin (Skin and subcutaneous tissue disorders) | 10 (15)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (18)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 1 (1)
electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
elevated LTF (Metabolism and nutrition disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
erectile dysfunction (Reproductive system and breast disorders) | 2 (3)
exostosis (Skin and subcutaneous tissue disorders) | 1 (1)
eye infection (Infections and infestations) | 2 (3)
fall (Injury, poisoning and procedural complications) | 1 (1)
fatigue (General disorders) | 26 (39)
febrile neutropenia (Infections and infestations) | 3 (3)
Fever (General disorders) | 7 (11)
flatulance (Gastrointestinal disorders) | 5 (5)
floater (Eye disorders) | 1 (2)
flu-like symptoms (General disorders) | 1 (1)
Flush (Vascular disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
fungal infection (Infections and infestations) | 8 (9)
aches (General disorders) | 1 (1)
hypergylcemia (Metabolism and nutrition disorders) | 27 (150)
hypoglymcemia (Metabolism and nutrition disorders) | 12 (30)
carpal tunel (Musculoskeletal and connective tissue disorders) | 1 (1)
hand tremors (Nervous system disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 11 (12)
heartburn (Gastrointestinal disorders) | 4 (4)
hematuria (Renal and urinary disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 32 (173)
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 (1)
herituism (Skin and subcutaneous tissue disorders) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
Hyperesthesia (Musculoskeletal and connective tissue disorders) | 1 (1)
hypertension (Vascular disorders) | 5 (5)
hypertochosis (Skin and subcutaneous tissue disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 22 (54)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin infection (Infections and infestations) | 5 (6)
sinus infection (Infections and infestations) | 1 (1)
finger infection (Infections and infestations) | 1 (1)
insomnia (Psychiatric disorders) | 12 (12)
itching (Skin and subcutaneous tissue disorders) | 1 (1)
IV infiltration (Skin and subcutaneous tissue disorders) | 1 (1)
karatoses (Skin and subcutaneous tissue disorders) | 1 (2)
kidney stone (Renal and urinary disorders) | 1 (1)
toe infection (Infections and infestations) | 1 (1)
leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
leg ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 23 (151)
light headedness (Nervous system disorders) | 1 (1)
loss of appetite (Metabolism and nutrition disorders) | 3 (3)
lymphopenia (Investigations) | 8 (79)
hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
mouth sores (Gastrointestinal disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 9 (16)
muscle cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 25 (35)
neutropenic fever (Blood and lymphatic system disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 4 (6)
night sweats (General disorders) | 4 (4)
numbness (Nervous system disorders) | 1 (1)
oral thrush (Infections and infestations) | 1 (1)
occular infection (Infections and infestations) | 1 (1)
hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
periorbital hair changes (Skin and subcutaneous tissue disorders) | 2 (2)
xerosis back (Skin and subcutaneous tissue disorders) | 1 (1)
buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
chest pain (General disorders) | 1 (2)
Hepatic pain (Hepatobiliary disorders) | 1 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Solar Plexis Pain (Nervous system disorders) | 1 (2)
forearm pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Upper Quadrant Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Scapula pain (Musculoskeletal and connective tissue disorders) | 1 (1)
stent pain (Injury, poisoning and procedural complications) | 1 (1)
palpitations (Cardiac disorders) | 4 (4)
paronychia (Infections and infestations) | 2 (5)
Pulmonary Embolism (Vascular disorders) | 4 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (20)
Platelet count decreased (Investigations) | 25 (81)
Pleural effusion (Reproductive system and breast disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
poison ivy (Skin and subcutaneous tissue disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 18 (58)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 3 (9)
rash (Skin and subcutaneous tissue disorders) | 33 (135)
rectal bleeding (Renal and urinary disorders) | 3 (3)
rectal fissure (Renal and urinary disorders) | 1 (1)
reflux (Gastrointestinal disorders) | 1 (2)
renal failure (Renal and urinary disorders) | 1 (1)
respiratory infection (Infections and infestations) | 1 (2)
rhinitis (Immune system disorders) | 2 (2)
rigors (General disorders) | 1 (1)
scratched cornea (Eye disorders) | 1 (1)
seasonal allergy (Immune system disorders) | 1 (1)
sepsis (Infections and infestations) | 3 (3)
septic shock (Infections and infestations) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (4)
sinus headache (Nervous system disorders) | 1 (1)
sinus tachcardia (Vascular disorders) | 1 (1)
sinusitus (Infections and infestations) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 23 (66)
somnolence (Nervous system disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
sweating (General disorders) | 3 (4)
syncope (Nervous system disorders) | 2 (2)
taste alteration (Gastrointestinal disorders) | 5 (5)
deep vein thrombosis (Vascular disorders) | 2 (2)
thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
thrombosis (Vascular disorders) | 2 (2)
thrush (Infections and infestations) | 4 (7)
trichomegaly (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
upset stomach (Gastrointestinal disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 4 (5)
vessel injury (Injury, poisoning and procedural complications) | 1 (1)
vomiting (Gastrointestinal disorders) | 14 (24)
weight loss (Investigations) | 10 (13)
yeast infection (Infections and infestations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes